CLINICAL TRIAL: NCT07038876
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy, Safety, and Tolerability of Orally Administered ML-007C-MA in Inpatient Adult Participants With Schizophrenia Experiencing an Acute Exacerbation of Psychosis
Brief Title: A Study to Assess the Efficacy and Safety of ML-007C-MA for the Treatment of Inpatient Adults With Schizophrenia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MapLight Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ML-007C-MA-211
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia
Keywords: Schizophrenia Spectrum and Other Psychotic Disorders Mental Disorders; Mental Disorders; Psychotic Disorders; Schizophrenia; Muscarinic Antagonists; Muscarinic Agonists; Cholinergic Agents
MeSH Terms: conditions — Schizophrenia; Mental Disorders; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- ML-007C-MA 330/6 mg QD (Experimental)
  Interventions: Drug: ML-007C-MA QD
- ML-007C-MA 210/3 mg BID (Experimental)
  Interventions: Drug: ML-007C-MA BID
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Matched Placebo
  Arms: Placebo
Drug: ML-007C-MA BID — ML-007C-MA dosed as 210/3 mg BID
  Arms: ML-007C-MA 210/3 mg BID
Drug: ML-007C-MA QD — ML-007C-MA dosed as 330/6 mg QD
  Arms: ML-007C-MA 330/6 mg QD

SUMMARY:
ML-007C-MA-211 is a Phase 2, randomized, double-blind, placebo-controlled study to evaluate the efficacy, safety, and tolerability of orally administered ML-007C-MA in inpatient adult participants aged 18 to 64 years with schizophrenia experiencing an acute exacerbation of psychosis.

The primary objective is to evaluate the efficacy of ML-007C-MA compared with placebo in the treatment of subjects with inadequately controlled symptoms of schizophrenia as measured by the Positive and Negative Syndrome Scale (PANSS) Total Score.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant has a primary diagnosis of schizophrenia based on the DSM-5 criteria that is confirmed by semi-structured clinical interview (Mini International Neuropsychiatric Interview for DSM-5).
* Participant may benefit from hospitalization or is currently hospitalized due to an acute exacerbation of schizophrenia symptoms, with exacerbation onset within 2 months of Screening. If the participant is already hospitalized for acute exacerbation of schizophrenia at Screening, they must have been inpatient for less than 2 weeks at the start of Screening.
* At Screening and Baseline, schizophrenia symptoms are at least moderate in severity and persistent, as defined by the PANSS and CGI-S.
* Participant is willing and able to be confined to an inpatient setting for the study duration, follow instructions, and adhere to protocol requirements.

Key Exclusion Criteria:

* Participant has any DSM-5 disorder, other than schizophrenia, within 12 months before Screening that is primarily responsible for the current symptoms or functional impairment.
* Participant has any psychiatric hospitalization(s) for more than 30 days (cumulative) during the 90 days before Screening and/or current involuntary hospitalization or incarceration.
* Participant received any antipsychotic medication or prohibited therapy within the Screening Period unless discontinued before Baseline.
* Participant has current evidence of a clinically significant and/or unstable medical comorbidity at Screening or Baseline.
* Participant is at an elevated risk of suicidal behavior.
* Participant has a known or likely allergy or other intolerance to ML-007C-MA, its active ingredients or their excipients or has a known or likely severe allergic reaction (eg, anaphylactic reaction, angioedema) to any drug that could pose a risk to the participant in this study.
* Participant has a DSM-5 diagnosis of moderate to severe substance use disorder (except tobacco or caffeine use disorder) within the 12 months before Screening (confirmed using Mini International Neuropsychiatric Interview).
* Participation in a clinical research study involving the administration of an investigational or marketed drug, biological product, or device within 90 days of Baseline, or concomitant active participation in an investigational study involving no drug, biological product, or device. Participants who have previously participated in a study with ML-007 may not participate.
* Participant is at elevated risk of violent or destructive behavior based on participant history and investigator judgment.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline to End of Treatment in Positive and Negative Syndrome Scale (PANSS) Total Score | Baseline and End of Treatment (5 weeks)
  The PANSS is a medical scale used for measuring symptom severity of participants with schizophrenia. The PANSS rating form contains 7 positive symptom scales, 7 negative system scales, and 16 general psychopathology symptom scales. Participants are rated from 1 to 7 on each symptom scale. The total score is the sum of all scales with a minimum score of 30 and a maximum score of 210. A decrease in PANSS total score correlates with an improvement in schizophrenia symptoms.

SECONDARY OUTCOMES:
Change From Baseline to End of Treatment in CGI-S score | Baseline and End of Treatment (5 weeks)
  The CGI-S is a clinician-rated assessment of the severity of a participant's current illness on a 7-point scale, where a higher score is associated with greater severity. Values range from 1 (not ill at all) to 7 (among the most extremely ill).
Change From Baseline to End of Treatment in PANSS-Marder positive factor score | Baseline and End of Treatment (5 weeks)
  The Positive Marder Factor score is derived from the PANSS and consists of the sum of 4 positive symptom items (P), one negative symptom item (N) and 3 general symptom items (G) (P1. Delusions; P3. Hallucinations; P5. Grandiosity; P6. Suspiciousness and persecution; N7. Stereotyped thinking; G1. Somatic concern; G9. Unusual thought content; G12. Lack of judgment and insight).
Change From Baseline to End of Treatment in PANSS-Marder negative factor score | Baseline and End of Treatment (5 weeks)
  The Negative Marder Factor score is derived from the PANSS and consists of the sum of 5 negative symptom items (N) and 2 general symptom items (G) (N1. Blunted affect; N2. Emotional withdrawal; N3. Poor rapport; N4. Passive/apathetic social withdrawal; N6. Lack of spontaneity; G7. Motor retardation; and G16. Active social avoidance), with a minimum score of 7 and a maximum score of 49.

CONTACTS AND LOCATIONS:
Overall Officials: MapLight Therapeutics, Study Director — MapLight Therapeutics
Locations (25):
- United States (25):
  - Clinical Site, Little Rock, Arkansas
  - Clinical Site, Bellflower, California
  - Clinical Site, Culver City, California
  - Clinical Site, Garden Grove, California
  - Clinical Site, Lemon Grove, California
  - Clinical Site, Los Angeles, California
  - Clinical Site, Montclair, California
  - Clinical Site, Orange, California
  - Clinical Site, Riverside, California
  - Clinical Site, San Diego, California
  - Clinical Site, Santee, California
  - Clinical Site, Sherman Oaks, California
  - Clinical Site, Torrance, California
  - Clinical Site, Hollywood, Florida
  - Clinical Site, Miami Lakes, Florida
  - Clinical Site, West Palm Beach, Florida
  - Clinical Site, Atlanta, Georgia
  - Clinical Site, Decatur, Georgia
  - Clinical Site, Chicago, Illinois
  - Clinical Site, Marlton, New Jersey
  - Clinical Site, Staten Island, New York
  - Clinical Site, North Canton, Ohio
  - Clinical Site, Austin, Texas
  - Clinical Site, DeSoto, Texas
  - Clinical Site, Richardson, Texas

IPD SHARING:
Plan to Share IPD: No